CLINICAL TRIAL: NCT03834272
Title: Feasibility of the LUM Imaging System for Detection of Peritoneal Surface Malignancies
Brief Title: Feasibility of the LUM Imaging System for Peritoneal Surface Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lumicell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLP-00010
Record Dates: First submitted 2019-02-04; First posted 2019-02-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-08

CONDITIONS: Peritoneal Metastases
Keywords: Gastrointestinal Cancer; Ovarian Cancer; Mesothelioma; Peritoneal surface malignancies
MeSH Terms: conditions — Gastrointestinal Neoplasms; Ovarian Neoplasms; Mesothelioma; Peritoneal Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- 1st Tier Dose Level- LUM Imaging System (Experimental): 3 patients will be administered a single dose of LUM015 at 1.0 mg/kg. Imaging with the LUM imaging device will be performed in vivo on surgical tissue.
  Interventions: Combination Product: LUM Imaging System
- 2nd Tier Dose Level- LUM Imaging System (Experimental): 9 patients will be administered a single dose of LUM015 at 1.5 mg/kg. Imaging with the LUM imaging device will be performed in vivo on surgical tissue. Some patients may be imaged with an additional imaging device.
  Interventions: Combination Product: LUM Imaging System
- 3rd Tier Dose Level- LUM Imaging System (Experimental): 6 patients will be administered a single dose of LUM015 at 2.0 mg/kg. Imaging with the LUM imaging device will be performed in vivo on surgical tissue. Some patients may be imaged with an additional imaging device.
  Interventions: Combination Product: LUM Imaging System

INTERVENTIONS:
Combination Product: LUM Imaging System — Patients will be injected with one of 3 study doses of LUM015 and tissue will be imaged in vivo with the LUM imaging device. Some patients may be imaged with an additional imaging device.

SUMMARY:
The objective of this feasibility study is to assess the initial safety and efficacy of the LUM Imaging System for in vivo imaging of metastases to the peritoneum from primary gastrointestinal cancer, ovarian cancer and mesothelioma. This feasibility study consists of a dose escalation phase to select the optimal dose.

DETAILED DESCRIPTION:
Subjects will be recruited and screened at a single institution, Massachusetts General Hospital. All subjects will have an established diagnosis of metastases to the peritoneum from primary colonic, appendiceal, or ovarian cancer or mesothelioma and are scheduled for surgical debulking. This study consists of a dose escalation and imaging timepoint evaluation.

18 patients will be enrolled into this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed metastases to the peritoneum from gastrointestinal cancer, ovarian cancer or mesothelioma prior to surgery.
* Subjects must be scheduled for surgical resection.
* Age of 18 years or older.
* Subjects must be able and willing to follow study procedures and instructions.
* Subjects must have received and signed an informed consent form.
* Subjects must be otherwise healthy except for the diagnosis of cancer, as per the criteria listed below.
* Subjects must have normal organ and marrow function as defined as:

  * Leukocytes > 3,000/mcL
  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Subjects with ECOG performance status of 0 or 1.

Exclusion Criteria:

* Subjects who are pregnant or nursing at the time of diagnosis.
* Subjects who are sexually active and not willing/able to use medically acceptable forms of contraception (hormonal or barrier method of birth control, abstinence) upon entering the study and for 60 days after injection of LUM015.
* Subjects who have taken an investigational drug within 30 days of enrollment.
* Subjects who have not recovered from adverse events due to other pharmaceutical or diagnostic agents.
* Subjects with uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 100 mm Hg; those subjects with known HTN should be under these values while under pharmaceutical therapy.
* History of allergic reaction attributed to drugs containing polyethylene glycol (PEG).
* History of allergic reaction to any oral or intravenous contrast agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, COPD or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive individuals on combination antiretroviral therapy are ineligible.
* Any subject for whom the investigator feels participation is not in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Initial efficacy of LUM015 in labeling peritoneal surface malignancies by molecular imaging by comparing imaging results with pathology | 1 Day
  Correlate the fluorescence levels in tumor tissue imaging to the dose of LUM015 injected.

SECONDARY OUTCOMES:
Number of patients with reported adverse events | up to 5 weeks post surgery
  Reported adverse events will be assessed and aggregated according to event type, relation to device or drug, and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Greer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No